CLINICAL TRIAL: NCT03835585
Title: The Provision of Gun Locks in Lethal Means Counseling to Increase Firearm Safety in a Suicide Risk Sample
Brief Title: Gun Locks in Firearm Suicide Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC#: 2018.26057
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Experimental group and comparison group measured immediately prior to intervention, immediately after intervention, 2 weeks after intervention, and one month after intervention. Analyses conducted will be Repeated Measures Analysis of Variance (RM-ANOVA).
Masking Description: Participants are informed that the purpose of the study is to "test the effects that providing gun locks as part of a psychological intervention has on gun safety behaviors" and that there are two treatment groups and that one is a "gun lock" group and that one is "standard intervention" group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gun lock (Experimental): Participants will be provided a gun lock and video instructions for its proper use, in addition to standard suicide risk interventions (i.e., standardized full suicide risk assessment, safety planning, lethal means counseling).
  Interventions: Device: Gun lock; Other: Suicide Risk Assessment; Behavioral: Safety Planning; Behavioral: Lethal Means Counseling
- Standard intervention (Active Comparator): Participants will be provided standard suicide risk interventions (i.e., standardized full suicide risk assessment, safety planning, lethal means counseling) without a gun lock. A gun lock and video instructions will be provided upon completion of the study.
  Interventions: Other: Suicide Risk Assessment; Behavioral: Safety Planning; Behavioral: Lethal Means Counseling

INTERVENTIONS:
Device: Gun lock — A cable-style gun lock that can be applied to a wide variety of guns for safe storage. The application of this device to most firearms renders them impossible to use properly while the device is in place and locked.
  Arms: Gun lock
Other: Suicide Risk Assessment — Thorough suicide risk assessment according to guidelines established by research (Joiner et al., 1999; Chu et al., 2015). This is used to determine the severity of suicide risk and appropriate actions to be taken.
Behavioral: Safety Planning — A psychological intervention for suicide risk that is based on research (Chu et al., 2015; Stanley & Brown, 2012). This involves listing the following on an index card: activities individuals can use to feel better during a crisis, contact numbers that are important to the individuals, emergency options that are always accessible, and reasons for living. Although the individualized nature of safety plans does not allow for a scripted/uniform approach, for this study they will all include 8 steps and steps 5-8 (emergency options) will be the same for each individual.
Behavioral: Lethal Means Counseling — A psychological intervention for suicide risk that is based on research (Bryan et al., 2011; Chu et al., 2015; Rudd, 2006; Stanley, 2018). This involves a psychological clinician discussing, with an at-risk individual, the importance for increasing the distance/obstacles between the individual at risk for suicide and specific types of lethal means. In the present study, the lethal means targeted was firearms and the lethal means counseling approach was able to be standardized/scripted as has been done in previous research (see Stanley, 2018).

SUMMARY:
This study compares the effectiveness of two interventions for suicide over the course of a month. The experimental intervention includes the provision of a gun lock with video instructions, in addition to standard suicide risk interventions (i.e., standardized full suicide risk assessment, safety planning, and lethal means counseling). The comparison intervention group will receive the same standard suicide risk interventions without the gun lock and video. The targeted outcome will be level of engagement in gun safety behaviors (e.g., using a gun lock, using a gun safe, considering getting rid of guns). It is predicted that the experimental intervention will result in greater increases over time in engagement in gun safety behaviors, as compared to the comparison intervention.

DETAILED DESCRIPTION:
Purpose: While psychology research and the suicide literature have not provided this evidence in a manner relevant to lethal means counseling, research across various disciplines has clearly demonstrated that providing individuals with gun locks and knowledgeable information about their proper use will significantly increase the likelihood that individuals will engage in firearm safety behaviors. The present study seeks to examine if the provision of gun locks, in addition to the current best standard interventions for suicide risk according to research, will significantly increase engagement in these behavioral outcomes.

Research Design/Method: The present study will utilize an experimental design with two groups, an experimental intervention group and a comparison intervention group. The experimental intervention group will receive the highest standard interventions (i.e., standardized full suicide risk assessment, safety planning, and lethal means counseling) in addition to a gun lock and instructional video. The comparison intervention group will receive the highest standard interventions, but will not be provided gun locks until after the study is complete.

The gun locks will be 15-inch cable locks. Locks will be mailed via USPS in envelopes upon completion of screener, if eligible for the study, but before they are scheduled to complete the first portion of the study. this will be arranged by making scheduling calls for initial sessions the day of/day after (depending on time) screeners are completed, scheduling initial sessions at least a week and a half after scheduling calls, and mailing the locks the day of scheduling calls.

Gun locks will be mailed to participants in the experimental intervention group. Data will be collected over three sessions. The first will be when baseline measures (e.g., demographics, outcomes) will be administered online, the intervention will be provided for all individuals by phone and online(only for the video instructions for lock), and post-intervention measures of outcome variables will assessed online. The 2-week follow-up interval and the 1-month interval will involve only assessment of the outcomes online. Participants in comparison intervention group will be provided gun locks after participation in the study is complete.

Research Question: Will the experimental intervention group outperform the comparison intervention group, regarding effectiveness in increasing engagement in firearm safety behaviors?

Hypothesis: The intervention for the experimental intervention group will be significantly more effective at increasing engagement in firearm safety behavior than that which will be provided for the comparison intervention group.

Data Analysis: Repeated Measures Analysis of Variance (RM-ANOVA) will be conducted, with a focus on measuring the interaction effects of Group and Time to assess whether experimental intervention group was significantly more effective than the comparison intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Must own and have access to a firearm
* Must have at least one lifetime episode of suicide ideation
* Must be 18 years of age or older

Exclusion Criteria:

- May not be under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
Engagement in Firearm Safety Behaviors | Immediately prior to intervention
  This includes a variety of actions and thinking patterns that promote safety regarding firearms. This is measured by a self-report instrument (Engagement in Firearm Safety Behaviors; Stanley, 2018), which contains 34 items. The items are scored on a Likert scale (i.e., 0 = Never; 1 = Sometimes, 2 = Often, 3 = Always) to gauge frequency of engagement. 16 items represent behaviors (e.g., "using a gun lock," "trading in your guns") and 18 represent thoughts (e.g., "thought about obtaining a gun lock," "thought about storing your gun unloaded.")
Engagement in Firearm Safety Behaviors | Two weeks after intervention
  This includes a variety of actions and thinking patterns that promote safety regarding firearms. This is measured by a self-report instrument (Engagement in Firearm Safety Behaviors; Stanley, 2018), which contains 34 items. The items are scored on a Likert scale (i.e., 0 = Never; 1 = Sometimes, 2 = Often, 3 = Always) to gauge frequency of engagement. 16 items represent behaviors (e.g., "using a gun lock," "trading in your guns") and 18 represent thoughts (e.g., "thought about obtaining a gun lock," "thought about storing your gun unloaded.")
Engagement in Firearm Safety Behaviors | One month after intervention
  This includes a variety of actions and thinking patterns that promote safety regarding firearms. This is measured by a self-report instrument (Engagement in Firearm Safety Behaviors; Stanley, 2018), which contains 34 items. The items are scored on a Likert scale (i.e., 0 = Never; 1 = Sometimes, 2 = Often, 3 = Always) to gauge frequency of engagement. 16 items represent behaviors (e.g., "using a gun lock," "trading in your guns") and 18 represent thoughts (e.g., "thought about obtaining a gun lock," "thought about storing your gun unloaded.")

SECONDARY OUTCOMES:
Intentions to Adhere to Clinician Recommendations | Immediately prior to Intervention
  A structured self-report questionnaire utilized in previous research (Stanley et al., 2017; Stanley, 2018) will be used in the present study to assess participants' intentions to adhere to clinician recommendations to limit access to a firearm for safety purposes. The two items will be rated on a 10-point Likert type scale (1 = Not At All Likely; 10 = Very Likely) and they will read as follows: 1) "How likely would you be to adhere to your clinician's recommendations to limit your access to a firearm for safety purposes?"; and 2) "How likely would you be to encourage a loved one to adhere to your clinician's recommendations to limit their access to a firearm for safety purposes?"
Intentions to Adhere to Clinician Recommendations | Immediately after intervention
  A structured self-report questionnaire utilized in previous research (Stanley et al., 2017; Stanley, 2018) will be used in the present study to assess participants' intentions to adhere to clinician recommendations to limit access to a firearm for safety purposes. The two items will be rated on a 10-point Likert type scale (1 = Not At All Likely; 10 = Very Likely) and they will read as follows: 1) "How likely would you be to adhere to your clinician's recommendations to limit your access to a firearm for safety purposes?"; and 2) "How likely would you be to encourage a loved one to adhere to your clinician's recommendations to limit their access to a firearm for safety purposes?"
Intentions to Adhere to Clinician Recommendations | Two weeks after intervention
  A structured self-report questionnaire utilized in previous research (Stanley et al., 2017; Stanley, 2018) will be used in the present study to assess participants' intentions to adhere to clinician recommendations to limit access to a firearm for safety purposes. The two items will be rated on a 10-point Likert type scale (1 = Not At All Likely; 10 = Very Likely) and they will read as follows: 1) "How likely would you be to adhere to your clinician's recommendations to limit your access to a firearm for safety purposes?"; and 2) "How likely would you be to encourage a loved one to adhere to your clinician's recommendations to limit their access to a firearm for safety purposes?"
Intentions to Adhere to Clinician Recommendations | One month after intervention
  A structured self-report questionnaire utilized in previous research (Stanley et al., 2017; Stanley, 2018) will be used in the present study to assess participants' intentions to adhere to clinician recommendations to limit access to a firearm for safety purposes. The two items will be rated on a 10-point Likert type scale (1 = Not At All Likely; 10 = Very Likely) and they will read as follows: 1) "How likely would you be to adhere to your clinician's recommendations to limit your access to a firearm for safety purposes?"; and 2) "How likely would you be to encourage a loved one to adhere to your clinician's recommendations to limit their access to a firearm for safety purposes?"
Acceptability of Intervention | Immediately prior to intervention
  The acceptability of the intervention will be measured utilizing the Client Satisfaction Questionnaire-8 (CSQ-8). The CSQ-8 is an 8-item instrument assessing the degree to which individuals find services to be acceptable (Attkisson & Zwick, 1982; Larsen et al., 1979). Items are rated in Likert type scales ranging from 1 to 4 (e.g., 1 = Quite dissatisfied, 2 = indifferent or mildly dissatisfied, 3 = Mostly satisfied, 4 = Very satisfied). The measure utilizes a summed score (range: 8-32), with higher values being indicative of higher levels of acceptability for the services received by respondents. Items cover a broad array of acceptability standards (e.g., "How satisfied are you with the amount of help you received?", "Have the services you received helped you to deal more effectively with your problems?").
Acceptability of Intervention | Immediately after intervention
  The acceptability of the intervention will be measured utilizing the Client Satisfaction Questionnaire-8 (CSQ-8). The CSQ-8 is an 8-item instrument assessing the degree to which individuals find services to be acceptable (Attkisson & Zwick, 1982; Larsen et al., 1979). Items are rated in Likert type scales ranging from 1 to 4 (e.g., 1 = Quite dissatisfied, 2 = indifferent or mildly dissatisfied, 3 = Mostly satisfied, 4 = Very satisfied). The measure utilizes a summed score (range: 8-32), with higher values being indicative of higher levels of acceptability for the services received by respondents. Items cover a broad array of acceptability standards (e.g., "How satisfied are you with the amount of help you received?", "Have the services you received helped you to deal more effectively with your problems?").
Acceptability of Intervention | Two weeks after intervention
  The acceptability of the intervention will be measured utilizing the Client Satisfaction Questionnaire-8 (CSQ-8). The CSQ-8 is an 8-item instrument assessing the degree to which individuals find services to be acceptable (Attkisson & Zwick, 1982; Larsen et al., 1979). Items are rated in Likert type scales ranging from 1 to 4 (e.g., 1 = Quite dissatisfied, 2 = indifferent or mildly dissatisfied, 3 = Mostly satisfied, 4 = Very satisfied). The measure utilizes a summed score (range: 8-32), with higher values being indicative of higher levels of acceptability for the services received by respondents. Items cover a broad array of acceptability standards (e.g., "How satisfied are you with the amount of help you received?", "Have the services you received helped you to deal more effectively with your problems?").
Acceptability of Intervention | One month after intervention
  The acceptability of the intervention will be measured utilizing the Client Satisfaction Questionnaire-8 (CSQ-8). The CSQ-8 is an 8-item instrument assessing the degree to which individuals find services to be acceptable (Attkisson & Zwick, 1982; Larsen et al., 1979). Items are rated in Likert type scales ranging from 1 to 4 (e.g., 1 = Quite dissatisfied, 2 = indifferent or mildly dissatisfied, 3 = Mostly satisfied, 4 = Very satisfied). The measure utilizes a summed score (range: 8-32), with higher values being indicative of higher levels of acceptability for the services received by respondents. Items cover a broad array of acceptability standards (e.g., "How satisfied are you with the amount of help you received?", "Have the services you received helped you to deal more effectively with your problems?").

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Joiner, PhD, Study Director — Robert O. Lawton Distinguished Professor; Bruno Chiurliza, MS, Principal Investigator — Graduate Student
Locations (1):
- Florida State University, Tallahassee, Florida, United States